CLINICAL TRIAL: NCT01342614
Title: The Effect of Metformin on the Correlation Between Hyperinsulinemia and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Prof. LI Guangwei, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET140
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2005-11

CONDITIONS: Diabetes Mellitus; Essential Hypertension
Keywords: Hypertension; Insulin Resistance; Hyperinsulinemia; Metformin; Fosinopril
MeSH Terms: conditions — Diabetes Mellitus; Essential Hypertension; Hypertension; Insulin Resistance; Hyperinsulinism | interventions — Fosinopril; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosinopril group (Active Comparator): Fosinopril group received fosinopril, 10mg, once per day.
  Interventions: Drug: Fosinopril
- Metformin group (Experimental): Metformin group was treated with metformin hydrochloride, 500mg, three times per day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Fosinopril — Fosinopril group received fosinopril, 10mg, once per day.
  Arms: Fosinopril group
Drug: Metformin — Metformin group was treated with metformin hydrochloride, 500mg, three times per day
  Arms: Metformin group

SUMMARY:
The objective of this study is to investigate the effect of metformin on the correlation between hyperinsulinemia and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65 years of age, regardless of sex
* duration of hypertension was <5 years
* overweight or obesity, mild to moderate hypertension, receive no euglycemic agent or antiobesity drug

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement | 8 weeks